CLINICAL TRIAL: NCT01857167
Title: Effect of Omega-3 Fatty Acids on Insulin Sensitivity in Chinese Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DUOLI2013011
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes; Insulin Resistance
Keywords: omega-3 fatty acids; randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Fish Oil Supplementation (Experimental): Patients will receive fish oil capsules, at a dose of 4g/day. Each 1g capsule will contain 300mg of EPA and 200mg of DHA.
  Interventions: Dietary Supplement: Fish Oil Supplementation
- Flaxseed Oil Supplementation (Experimental): Patients will receive flaxseed oil capsule, at a dose of 4g/day. Each 1g capsule will contain 630mg of ALA
  Interventions: Dietary Supplement: Flaxseed Oil Supplementation
- Placebo Supplementation (Placebo Comparator): Patients will receive corn oil in the capsules at the same dose as fish oil. The corn oil will appear identical in size and color to the fish oil.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil Supplementation
  Arms: Fish Oil Supplementation
Dietary Supplement: Flaxseed Oil Supplementation
  Arms: Flaxseed Oil Supplementation
Dietary Supplement: placebo
  Arms: Placebo Supplementation

SUMMARY:
This study is to examine the change of fasting insulin, glucose, insulin sensitivity and related traits in response to the six month treatment of omega-3 fatty acids, including fish oil and flaxseed oil, in Chinese type 2 diabetic patients. Corn oil, rich in omega-6 fatty acids, will be selected as a controlled oil. The investigators hypothesize that omega-3 fatty acids could improve insulin sensitivity and glucose metabolism in Chinese type 2 diabetic patients.

DETAILED DESCRIPTION:
The insulin resistance will be estimated by a homeostatic model assessment model of insulin resistance (HOMA-IR)

ELIGIBILITY:
Inclusion Criteria:

1. Fasting glucose > 7.0 or have diabetes medication;
2. Male, 35-80 years; female, postmenopausal to 80 years;
3. Agree to participant in the trial.

Exclusion Criteria:

1. Deny to sign the informed consent;
2. type 1 diabetes;
3. Family history of hypertriglyceridemia or fasting triglyceride>4.56 mmol/L;
4. Have severe liver disease, kidney disease or cancer;
5. Participating in the other clinical trial within 30 days;
6. Other diseases or conditions, for which the doctor of the patients do not agree his or her participating.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Zheng JS, Huang T, Yang J, Fu YQ, Li D. Marine N-3 polyunsaturated fatty acids are inversely associated with risk of type 2 diabetes in Asians: a systematic review and meta-analysis. PLoS One. 2012;7(9):e44525. doi: 10.1371/journal.pone.0044525. Epub 2012 Sep 11. PMID 22984522
- [Derived] Zheng JS, Lin M, Fang L, Yu Y, Yuan L, Jin Y, Feng J, Wang L, Yang H, Chen W, Li D, Tang J, Cai W, Shi M, Li Z, Wang F, Li D. Effects of n-3 fatty acid supplements on glycemic traits in Chinese type 2 diabetic patients: A double-blind randomized controlled trial. Mol Nutr Food Res. 2016 Oct;60(10):2176-2184. doi: 10.1002/mnfr.201600230. Epub 2016 Jul 12. PMID 27279274